CLINICAL TRIAL: NCT05949073
Title: The Impact of Retraction Cords Used in Fixed Prosthodontics on the Gingival Margin Level in Humans: A Clinical Study.
Brief Title: The Impact of Retraction Cords on the Gingival Margin Level.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Majdoleen Fouad, Postgraduate Student., University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Retraction cords
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Gingival Retraction; Gingival Recession; Periodontal Health
Keywords: retraction cords; gingival recession; periodontal health; gingival retraction
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non impregnated gingival retraction cord - less than 10 minutes (Active Comparator): Non impregnated gingival retraction cord will be placed around the prepared tooth and left for less than 10 minutes.
  Interventions: Procedure: Non-impregnated retraction cords/ less than 10 minutes
- Non impregnated gingival retraction cord - more than 10 minutes (Active Comparator): Non impregnated gingival retraction cord will be placed around the prepared tooth and left for more than 10 minutes.
  Interventions: Procedure: Non-impregnated retraction cords/ more than 10 minutes
- impregnated gingival retraction cord - less than 10 minutes (Active Comparator): Impregnated gingival retraction cord will be placed around the prepared tooth and left for less than 10 minutes.
  Interventions: Drug: impregnated gingival retraction cord - less than 10 minutes
- impregnated gingival retraction cord - more than 10 minutes (Active Comparator): Impregnated gingival retraction cord will be placed around the prepared tooth and left for more than 10 minutes.
  Interventions: Drug: impregnated gingival retraction cord - more than 10 minutes

INTERVENTIONS:
Procedure: Non-impregnated retraction cords/ less than 10 minutes — lower first molar will be prepared for full coverage restoration, plain retraction cord will be placed in the sulcus just before impression recording (less than 10 minutes).
  Arms: Non impregnated gingival retraction cord - less than 10 minutes
Procedure: Non-impregnated retraction cords/ more than 10 minutes — the preparation of the lower first molar for full coverage restoration will be initiated - occlusal reduction, contact points breaking, and preparation with the roughest bur- then a plain retraction cord will be placed and kept in the sulcus until finishing the preparation and impression recording which will take more than 10 minutes.
  Arms: Non impregnated gingival retraction cord - more than 10 minutes
Drug: impregnated gingival retraction cord - less than 10 minutes — lower first molar will be prepared for full coverage restoration, Aluminum chloride-impregnated retraction cord will be placed in the sulcus just before impression recording (less than 10 minutes).
  Other Names: Aluminum chloride-impregnated retraction cords.
  Arms: impregnated gingival retraction cord - less than 10 minutes
Drug: impregnated gingival retraction cord - more than 10 minutes — the preparation of the lower first molar for full coverage restoration will be initiated - occlusal reduction, contact points breaking, and preparation with the roughest bur- then an Aluminum chloride-impregnated retraction cord will be placed and kept in the sulcus until finishing the preparation and impression recording which will take more than 10 minutes.
  Other Names: Aluminum chloride-impregnated retraction cord
  Arms: impregnated gingival retraction cord - more than 10 minutes

SUMMARY:
The purpose of this study is to examine the relationship between placing specific retraction cord for different periods of time and the post-operative gingival margin level in humans. Determining the amount of immediate reversible and delayed irreversible gingival recession (vertical gingival retraction) that might happen after placing a retraction cord around a natural tooth in healthy humans. It also aims to investigate the impact of mechanical and chemo-mechanical gingival retraction on periodontal health.

DETAILED DESCRIPTION:
Dental impression is the communication tool between the dentist and the dental technician during the fabrication of fixed dental prosthesis, capturing a precise impression of the prepared tooth and the finish line is mandatory to ensure the perfect fitting of the final prosthesis.

Atraumatic gingival displacement is performed to provide sufficient both lateral and vertical space between the finish line and the gingival tissue that will allow recording adequate amount of unprepared tooth structure with the least distortion of impression material as well as minimal damage to attachment apparatus of the tooth as maintaining a healthy periodontium is an important factor in the survival of any fixed prosthesis.

The gingival recession that might happen after soft tissue displacement may jeopardize treatment success in esthetic areas of the mouth. Knowledge about the soft tissue reaction to one of the most common gingival displacement methods (retraction cords) is critical yet limited. Also, there is a gap in knowledge about the safety of retraction cords when used for multiple teeth preparations and would then be left in the sulcus for an extended amount of time, as well as the potential harm they can do in terms of persistent gingival recession.

The purpose of this study is to examine the relationship between placing specific retraction cords for different periods of time and the post-operative gingival margin level in humans. Determining the amount of immediate reversible and delayed irreversible gingival recession (vertical gingival retraction) that might happen after placing a retraction cord around a natural tooth in healthy humans. It also aims to investigate the impact of mechanical and chemo-mechanical gingival retraction on periodontal health.

This clinical study is expected to be useful for dental clinicians who use retraction cords during restorative procedures (cervical composite restorations) or for fixed prostheses; awareness about the amount of transient and permanent gingival recession that could occur is important to avoid undesirable effects such as esthetic issues and/or sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-50 years
2. Systemically healthy no history of medical disease
3. Volunteers should have a lower first molar indicated for full coverage restoration, of healthy periodontium with an antagonist tooth and proximal contacts.
4. Gingival index score 0,1
5. Plaque index score 0,1
6. Probing depth ≤3 mm
7. No bleeding on probing.

Exclusion Criteria:

1. Gingival and periodontal disease
2. Pregnancy and lactation
3. History of systemic diseases such as hypertension, diabetes mellitus, HIV, bone metabolic disorders, radiation therapy, and cancer.
4. History of prolonged use of steroids/immunosuppressive agents/aspirin/anticoagulant/other medications.
5. Heavy Smoking.
6. Deleterious habits.
7. Teeth with high scalloped margins, keratinized tissue less than 2 mm, fibrotic gingival tissue, gingival recession, pocket formation deeper than 3mm.
8. Teeth with thick flat gingival phenotype.
9. Teeth with Sub-gingival caries or restoration at the buccal surface.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The amount of irreversible gingival recession that might happen after gingival retraction. | 4 weeks
  The amount of reversible and irreversible gingival recession (vertical gingival retraction) that might occur in healthy humans after placing retraction cords around prepared teeth for different periods of time. This will be measured after recording multiple digital intraoral scans pre-operative, 1 week, and 4 weeks post-operative using Medit i-700 then they will be superimposed using Medit Design tool (previously known as Medit compare) to track the vertical location of the gingival margin.

SECONDARY OUTCOMES:
The impact of retraction cords on periodontal health. | 4 weeks
  The impact on periodontal health will be measured by recording the periodontal indices pre-operative, 1-week, and 4 weeks post-operative by a single-blinded periodontist.
The level of patient's discomfort. | Immediately after the intervention
  The patient's level of discomfort will be recorded using the Numerical Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Mahmoud, Phd, Study Director — University of Jordan
Locations (1):
- the University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Hamad KQ, Azar WZ, Alwaeli HA, Said KN. A clinical study on the effects of cordless and conventional retraction techniques on the gingival and periodontal health. J Clin Periodontol. 2008 Dec;35(12):1053-8. doi: 10.1111/j.1600-051X.2008.01335.x. PMID 19040582
- [Background] Ruel J, Schuessler PJ, Malament K, Mori D. Effect of retraction procedures on the periodontium in humans. J Prosthet Dent. 1980 Nov;44(5):508-15. doi: 10.1016/0022-3913(80)90069-4. PMID 7003108
- [Background] Sarmento HR, Leite FR, Dantas RV, Ogliari FA, Demarco FF, Faot F. A double-blind randomised clinical trial of two techniques for gingival displacement. J Oral Rehabil. 2014 Apr;41(4):306-13. doi: 10.1111/joor.12142. Epub 2014 Jan 22. PMID 24446590
- [Background] Feng J, Aboyoussef H, Weiner S, Singh S, Jandinski J. The effect of gingival retraction procedures on periodontal indices and crevicular fluid cytokine levels: a pilot study. J Prosthodont. 2006 Mar-Apr;15(2):108-12. doi: 10.1111/j.1532-849X.2006.00083.x. PMID 16650011
- [Background] Einarsdottir ER, Lang NP, Aspelund T, Pjetursson BE. A multicenter randomized, controlled clinical trial comparing the use of displacement cords, an aluminum chloride paste, and a combination of paste and cords for tissue displacement. J Prosthet Dent. 2018 Jan;119(1):82-88. doi: 10.1016/j.prosdent.2017.03.010. Epub 2017 May 5. PMID 28478985